CLINICAL TRIAL: NCT01491269
Title: Guided Internet-delivered Cognitive-behavioral Therapy for Former Chronic Pain Patients: Randomised Controlled Trial
Brief Title: Guided Internet-delivered Cognitive-behavioral Therapy for Former Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerhard Andersson (Other Government)
Responsible Party: Sponsor-Investigator, Gerhard Andersson, professor, Linkoeping University, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: smartaMB2011
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain
Keywords: chronic pain; internet delivered CBT; tertiary intervention; mindfulness; applied relaxation; guided self help
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet delivered CBT (Experimental): Internet delivered cognitive behavioral intervention, 8 weeks treatment.
  Interventions: Behavioral: Guided Internet-based cognitive behavioural treatment
- No intervention (No Intervention): Waitlist

INTERVENTIONS:
Behavioral: Guided Internet-based cognitive behavioural treatment — Eight weeks internet-based cognitive behavioural treatment. Treatment consisted of education, cognitive skills acquisition, behavioural rehearsal, generalization and maintenance.
  Arms: Internet delivered CBT

SUMMARY:
The aim of the present study was to investigate if guided Internet-delivered Cognitive-behavioral Therapy (CBT) would help chronic pain patients who had previously undergone a multidisciplinary treatment but still have residual problems.

DETAILED DESCRIPTION:
The present study investigates Internet-delivered CBT as a tertiary intervention. This is motivated by the fact that many pain patients relapse after rehabilitation and some may be in need of additional treatment. The persons who fulfills the inclusion criteria undergoes a structured telephone interview. The study is a experimental design with a treatment and an active control group measured before and after a treatment period. The control group were invited to participate in a moderated online discussion forum. Follow up data was collected six months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* to have been medically investigated (within one year)
* completed the multidisciplinary rehabilitation program
* have residual symptoms after the rehabilitation treatment (defined as functional impairment caused by their pain)
* have Internet access

Exclusion Criteria:

* planned surgery
* ongoing medical investigation that could impede participation in the study
* suffering from acute physical or psychological conditions
* people confined to wheelchairs
* people not fluent with the Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The Coping Strategies Questionnaire (CSQ) | One week pre treatment, one week post treatment
  The CSQ contains 50 items divided in eight scales that measures different cognitive and behavioral coping strategies. The different coping strategies are: diverting attention, re-interpreting pain sensations, coping self-statements, ignoring sensations, praying and hoping, catastrophizing, increased behavioral activities and pain behavior (Rosenthiel & Keefe, 1983). Change from baseline in the different subscales pre- and post treatment.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale, HADS | One week pre treatment, one week post treatment
  HADS is a 14-item questionnaire, and is designed to measure anxiety and depression in non-psychiatric patients.
Multidimensional Pain Inventory, MPI | One week pre treatment, one week post treatment
  MPI, assess psychosocial and behavioural consequences of pain. It´s divided into 2 sections and consisting of 8 scales. These are: Pain Severity, Interference, Life Control, Affective Distress, Support, Punishing Responses, Solicitous Responses and Distracting Responses.
Pain and Impairment Relationship Scale (PAIRS) | One week pre treatment, one week post treatment
  PAIRS consist of 15 personal statements that reflect thoughts, attitudes and opinions about pain. The questionnaire assesses beliefs and attitudes that patients have regarding pain and ability to function despite discomfort.
Quality of Life Inventory (QOLI) | One week pre treatment, one week post after treatment
  QOLI contains 32 items for assessing life satisfaction. The assessment yields an overall score and profile in 16 areas of life; health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighborhood and community. Each item is rated in terms of importance and satisfaction.
Chronic Pain Acceptance Questionnaire (CPAQ) | One week pre treatment, one week post treatment
  CPAQ contains 20 items divided in two scales, engagement and willingness. CPAQ measures acceptance in relation to chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Study Director — Linkoeping University; Monica Buhrman, MSc, Principal Investigator — Uppsala University; Timo Hursti, PhD, Study Chair — Uppsala University; Torsten Gordh, Professor, Study Chair — Uppsala University; Anna Fredriksson, MSc, Study Chair — Uppsala University; Gunnel Edström, MSc, Study Chair — Uppsala University; Dorna Shaffi, MSc, Study Chair — Uppsala University; Carolina Törnqvist, MSc, Study Chair — Uppsala University; Brjann Ljotsson, PhD, Study Chair — Karolinska Institutet, Stockholm
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No